CLINICAL TRIAL: NCT06774898
Title: Spinal Bracing in Adults with Painful Degenerative Scoliosis: a Randomized Controlled Open Trial
Acronym: BRASCO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP230815
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Degenerative Scoliosis; Scoliosis Idiopathic; Thoracolumbar Scoliosis
Keywords: Scoliosis; Low back pain; Spine; Bracing
MeSH Terms: conditions — Scoliosis; Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A : A custom-molded lumbar-sacral orthosis (Experimental)
  Interventions: Device: Custom-molded lumbar-sacral orthosis; Other: Usual Care
- Arm B : a standardized prescription of 20 outpatient physiotherapy sessions (No Intervention)

INTERVENTIONS:
Device: Custom-molded lumbar-sacral orthosis — A custom-molded lumbar-sacral orthosis made according to the Vésinet method associated with measures designed to enhance adherence based on goal-setting techniques (i.e. personalized advice, self-determination of the wearing time, hotline) techniques and monitoring of adherence using a temperature sensor chip to provide feedbacks to participants on the wearing time at follow-up visits, and usual care (i.e. a standardized prescription of 20 outpatient physiotherapy sessions including active self-correction, spinal muscle strengthening, spine and lower limb stretching and learning of home-based exercises).
  Arms: Arm A : A custom-molded lumbar-sacral orthosis
Other: Usual Care — Usual care consisting in a standardized prescription of 20 outpatient physiotherapy sessions including active self-correction, spinal muscle strengthening, spine and lower limb stretching and learning of home-based exercises
  Arms: Arm A : A custom-molded lumbar-sacral orthosis

SUMMARY:
The purpose of this study is to compare the efficacy on low back pain intensity at 6 months after randomization of a custom-molded lumbar-sacral orthosis as an add-on therapy to usual care in people with painful adult degenerative scoliosis.

DETAILED DESCRIPTION:
Adult degenerative scoliosis is a spinal deformity that appears during adulthood, usually after 50 years, on a previous aligned spine or on an idiopathic scoliosis, due to a cascade of degenerative changes. Adult degenerative scoliosis is more prevalent in women than in men and affects up to 40% of adults aged 65 years and older. Overall, 60 to 80% of patients with adult degenerative scoliosis suffer from low back pain. Apart from analgesics, spinal glucocorticoid injections and physiotherapy, the 2 therapeutic options are bracing and spinal surgery.

Recent literature has suggested better outcomes with surgery than with conservative care. However, the level of evidence was low and the use of bracing in the conservative approach was not specifically evaluated. Therefore, good quality studies assessing bracing efficacy in adult degenerative scoliosis are lacking, explaining in part why many physicians do not offer it as a first-line therapeutic option and instead refer patients to surgery. In a retrospective study of 38 patients with adult degenerative scoliosis, the use of a custom-molded lumbar-sacral orthosis, for a minimum of 6h/d, was associated with a reduction in curve progression as measured with the Cobb angle and with an improvement in pain and activity limitations, at 5-year follow-up.

We hypothesize that a custom-molded lumbar-sacral orthosis as an add-on therapy to usual care (i.e. a standardized prescription of 20 outpatient physiotherapy sessions) could decrease symptoms in people with painful adult degenerative scoliosis as compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 to 75 years,
* Degenerative thoracolumbar or lumbar scoliosis with Cobb angle for the largest curve greater than 20°on EOS® full-spine X-ray less than 1 year (this can be a de-novo scoliosis, or a degenerative scoliosis that appears on an idiopathic scoliosis), and
* Low back pain with a duration more than 3 months
* Low back pain with an intensity greater than 40 of 100 points on a self-administered numeric rating scale.
* Patient able to give written informed consent prior to participation in the study Affiliation with a mode of social security (profit or being entitled).

Exclusion Criteria:

* Spinal deformity secondary to a specific condition (e.g. fracture, infection, tumour, inflammatory rheumatic disease, neuromuscular disorder, genetic disorder),
* History of spine surgery,
* Morphotype and/or conditions making spinal bracing technically impossible (e.g. obesity, severe clinical sagittal and/or coronal malalignment, recent abdominal surgery etc)
* Inability to speak and/or read French language,
* Inability or refusal to wear a custom-molded lumbar-sacral orthosis,
* Patients already wearing a custom-molded lumbar-sacral orthosis,
* Cognitive disorders,
* People under tutorship or curatorship,
* Protected adults, and
* Patients on AME (state medical aid),
* Pregnant women

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-02-02 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2029-02-02 (Estimated)

PRIMARY OUTCOMES:
Low back pain intensity | 6 months after randomization
  Mean variation from baseline in low back pain intensity at 6 months after randomization, using a self-adminitred 11-point numeric rating scale

SECONDARY OUTCOMES:
Low back pain intensity | 12 and 24 months after randomization
  Mean variation from baseline in low back pain intensity at 12 and 24 months after randomization, using a self-adminitred 11-point numeric rating scale (0, no pain and 100, maximal pain in 10-point increments)
Spine-specific activity limitations | 6,12 and 24 months
  Mean variation in spine-specific activity limitations using the self-administered Oswestry Disability Index (ODI, 0 no limitations and 100, maximal limitations) at 6, 12 and 24 months,
Health-related quality of life | 6,12 and 24 months
  Mean variation in health-related quality of life using the self-administered EQ-5D-5L questionnaire (1, having no problems and 5, having extreme problems) at 6, 12 and 24 months,
Progression of the lumbar curve | 12 and 24 months
  Percentage of participants with a progression of the lumbar curve, as measured by the Cobb angle, greater than 5° on an EOS® full-spine X-ray standardized posteroanterior X-ray in standing, weight-bearing position (EOS® full-spine X-ray system) at 12 and 24 months
Spine surgery | 24 months
  Percentage of participants who self-report spine surgery at 24 months
Cost-utility ratio | 24 months
  Estimated total costs and incremental cost-utility ratio at 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Service de Rééducation et de Réadaptation de l'Appareil Locomoteur et des Pathologies du Rachis, Hôpital Cochin, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No